CLINICAL TRIAL: NCT07320560
Title: Personalized Atrial Fibrillation Ablation Guided by Non-Invasive Global Mapping - the CURE-AF Pilot Study
Brief Title: Personalized Atrial Fibrillation Ablation Guided by Non-Invasive Global Mapping
Acronym: CURE-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Heart Institute (Other)
Responsible Party: Principal Investigator, Till Althoff, Head of Research and Principal Investigator, German Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA1/204/25
Record Dates: First submitted 2025-11-27; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Catheter Ablation; Non-invasive mapping; Global Mapping; Electrocardiographic Imaging; Body Surface Mapping; Atrial fibrillation drivers
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-invasive mapping-guided ablation (Experimental): In this arm patients undergo a personalized ablation approach: In addition to conventional pulmonary vein isolation, additional target regions will be ablated based on non-invasive global mapping.
  Interventions: Procedure: Non-invasive mapping-guided ablation

INTERVENTIONS:
Procedure: Non-invasive mapping-guided ablation — The study intervention consists of
  1. Empirical pulmonary vein isolation (current standard of care) plus
  2. A personalized ablation approach targeting up to three additional atrial regions which harbour critical AF-perpetuating sources:
     * Target regions are selected based on the temporal Stability of local Atrial High-Rate Activity (SAHRA) using a non-invasive global mapping system (Acorys, Corify Care). Local high-rate activity is confirmed by endocardial mapping.
     * Selected target regions displaying stable high-rate activity are isolated or homogenized according to predefined regional borders based on the 15-segment bi-atrial model of the EHRA and EACVI Clinical Consensus on Standardized Atrial Regionalization (Althoff et al. 2025).

SUMMARY:
This pilot study investigates if non-invasive global mapping can guide catheter ablation of atrial fibrillation (AF) by defining personalized targets based on the temporal Stability of local Atrial High-Rate Activity (SAHRA). The study also assesses efficacy and safety of this approach and evaluates potential signals of harm. The main questions it aims to answer are:

* Does ablation of targets defined by non-invasive global mapping improve rates of acute atrial fibrillation termination?
* Does such a personalized ablation approach reduce arrhythmia recurrence rates? Researchers will compare the results of the personalized ablation approach with comparable patients that had undergone a conventional "empirical" ablation approach (pulmonary vein isolation).

Participants will:

* Undergo a personalized catheter ablation approach employing both a non-invasive global mapping system and a conventional intracardiac mapping system
* Visit the clinic 3, 6 and 12 months after ablation for clinical follow-up
* Schedule a telephone visit 9 and 24 months after ablation for clinical follow-up

DETAILED DESCRIPTION:
The aim of this study is to test the feasibility and potential of a personalized, non-invasive mapping-guided ablation approach in patients with persistent atrial fibrillation (AF), who are unlikely to benefit from empirical pulmonary vein isolation alone. As a pilot study, it is designed to assess feasibility and procedural efficacy as well as potential signals of harm.

General Strategy:

Patients with persistent AF planned for catheter ablation are eligible in case of left atrial enlargement.

The study intervention consists of two steps:

1. Empirical pulmonary vein isolation in all patients (current standard of care).
2. A personalized ablation approach targeting up to three additional atrial regions which harbour critical AF-perpetuating sources:

   * Target regions are selected based on the temporal Stability of local Atrial High-Rate Activity (SAHRA) using a non-invasive global mapping system (Acorys, Corify Care).
   * Selected target regions displaying stable high-rate activity are isolated or homogenized according to predefined regional borders based on the 15-segment bi-atrial model of the EHRA and EACVI Clinical Consensus on Standardized Atrial Regionalization.

ELIGIBILITY:
Inclusion Criteria:

Ablation-naïve patients with:

1. Persistent AF planned for catheter ablation plus
2. Left atrial enlargement (LA diameter ≥45 mm or LA volume index ≥35ml/m2 or LA area ≥20 cm2)

Exclusion Criteria:

* Previous cardiac ablation
* Age <18 years
* Pregnancy or lactation
* Previous stroke/TIA
* Severe left ventricular dysfunction (LVEF <35%)
* Renal failure (GFR <30 ml/min)
* Dermal disease or hypersensitivity predisposing for skin irritation or exanthema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of acute AF termination | Procedural
  Acute AF termination (to sinus rhythm or conversion into an organized atrial tachycardia) upon ablation

SECONDARY OUTCOMES:
Proportion of patients with arrhythmia-free survival | Days 91 to 365 post-ablation
  Absence of any atrial tachyarrhythmia (atrial fibrillation [AF], atrial flutter [AFL] or atrial tachycardia [AT]) between days 91 and 365 post ablation. AF, AFL or AT will qualify as a recurrence after ablation if it lasts 30 s or longer.
Proportion of patients with AF-free survival | Days 91 to 365 post-ablation
  Absence of atrial fibrillation [AF] between days 91 and 365 post ablation. AF will qualify as a recurrence after ablation if it lasts 30 s or longer.
Time to arrhythmia recurrence | Days 91 to 365 post-ablation
  Time to first atrial tachyarrhythmia (atrial fibrillation [AF], atrial flutter [AFL] or atrial tachycardia [AT]) between days 91 and 365 post ablation. AF, AFL or AT will qualify as a recurrence after ablation if it lasts 30 s or longer.
Time to AF recurrence | Days 91 to 365 post-ablation
  Time to first atrial fibrillation [AF] between days 91 and 365 post ablation. AF will qualify as a recurrence after ablation if it lasts 30 s or longer.
Rate of procedure-related complications | Day 0 to 30 post-ablation
  Composite safety endpoint composed of:
  * cardiac tamponade requiring drainage
  * persistent phrenic nerve palsy lasting >24 hours
  * serious vascular complications requiring intervention
  * stroke/TIA
  * atrioesophageal fistula
  * death

OTHER OUTCOMES:
Procedure time | Day 0
  Skin-to-skin duration of the ablation (procedural endpoint)
Total left atrium indwelling time | Day 0
  Procedural endpoint
Fluoroscopy time | Day 0
  Procedural endpoint
Hemolysis marker levels on day 1 post-ablation | Day 1 post-ablation
  Procedural endpoint
GFR on day 1 post-ablation | Day 1 post-ablation
  Procedural endpoint
Proportion of patients with acute renal failure | Day 0 to 30 post-ablation
  Procedural endpoint
hsTroponin on day 1 post-ablation | Day 1 post-ablation
  Procedural endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Till F Althoff, M.D., Principal Investigator — German Heart Center of the Charitè, Berlin, Department of Cardiology, Angiology and Intensive Care Medicine
Locations (5):
- Germany (2):
  - German Heart Center of the Charité, Charité University Hospital Berlin, Berlin
  - Frankfurt University Heart and Vascular Center, Frankfurt am Main
- Central Lisbon University Hospital Centre (CHULC), Hospital de Santa Marta, Lisbon, Portugal
- Spain (2):
  - Hospital Clinic, University of Barcelona, Barcelona
  - Gregorio Marañón General University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: No
Data underlying published results will be provided upon reasonable request

REFERENCES:
- [Background] Invers-Rubio E, Hernandez-Romero I, Reventos-Presmanes J, Ferro E, Guichard JB, Regany-Closa M, Pellicer-Sendra B, Borras R, Prat-Gonzalez S, Tolosana JM, Porta-Sanchez A, Arbelo E, Guasch E, Sitges M, Brugada J, Guillem MS, Roca-Luque I, Climent AM, Mont L, Althoff TF. Regional conduction velocities determined by noninvasive mapping are associated with arrhythmia-free survival after atrial fibrillation ablation. Heart Rhythm. 2024 Sep;21(9):1570-1580. doi: 10.1016/j.hrthm.2024.04.063. Epub 2024 Apr 16. PMID 38636930
- [Background] Althoff TF, Anderson RH, Goetz C, Petersen SE, Diaz PM, Nijveldt R, Maurovich-Horvat P, Bax J, Hussain S, Schmidt C, Spicer DE, Sanchez-Quintana D, Corsi C, Dossel O, Climent AM, Rodriguez B, Schotten U, Loewe A, Guillem MS, Cabrera JA, Merino JL, Wijnmaalen AP, Bertrand PB, de Groot N, Derval N, Didenko M, Donal E, Dweck MR, Ho SY. Regionalization of the atria for 3D electroanatomical mapping, cardiac imaging, and computational modelling: a clinical consensus statement of the European Heart Rhythm Association and the European Association of Cardiovascular Imaging of the ESC. Europace. 2025 Jul 1;27(7):euaf134. doi: 10.1093/europace/euaf134. PMID 40736086